CLINICAL TRIAL: NCT01736943
Title: Phase II Trial of the Combination of Subcutaneous (SQ) Bortezomib and Pegylated Liposomal Doxorubicin (PLD or Doxil or LipoDox) for the Treatment of Patients With Relapsed/Refractory Acute Myelogenous Leukemia (AML)
Brief Title: Bortezomib and Doxil for the Treatment of Patients With Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph Tuscano (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Joseph Tuscano, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 322070; UCDCC#230 (Other: UC Davis); X05385 (Other Grant/Funding Number: Millennium Pharmaceuticals)
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Bortezomib; Doxil
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Bortezomib; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib + Doxil (Experimental): Bortezomib will be given subcutaneously at 1.5mg/m2 on days 1, 4, 8 and 11 of a 3 week cycle. Doxil will be administered once every three weeks as a single intravenous infusion at a dose of 40 mg/m2 (day 4 of each cycle).
  Interventions: Drug: Bortezomib; Drug: Doxil

INTERVENTIONS:
Drug: Bortezomib — Bortezomib will be given twice a week subcutaneously (under the skin) for two weeks in every 3 week cycle.
  Other Names: Velcade
Drug: Doxil — Doxil or LipoDox will also be given through a venous catheter (inside your vein). Doxil or LipoDox will be given over 60 to 90 minutes on Day 4 of every 21-day cycle.
  Other Names: LipoDox; pegylated liposomal doxorubicin

SUMMARY:
The purpose of this study is to determine whether bortezomib in combination with doxil/lipodox is effective in the treatment of Acute Myeloid Leukemia.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) remains largely incurable despite advances that have been made in recent years into increasing the complete response (CR) rates. In elderly patients (over the age of 60), CR rates are lower, 40 to 50%, and long term disease-free and overall survival is less than 10%. The therapeutic options for relapsed/refractory AML are significantly limited. Bortezomib has shown promising activity in patients with advanced hematologic malignancies, including those with leukemia and non-Hodgkin's lymphoma.

Given the available data suggesting efficacy of bortezomib in combination with doxil in patients with relapsed multiple myeloma (MM), chronic lymphocytic leukemia (CLL), and Non Hodgkin's lymphoma (NHL) as well as the known sensitivity of AML to anthracyclines and in vitro data demonstrating the sensitivity of multiply resistant AML cells to bortezomib, we are proposing the use of this combination in patients with relapsed/refractory AML or elderly patients who are not candidates for standard induction therapy.

Using the subcutaneous formulation of bortezomib would provide patients with reduced neurotoxicity and easier schedule due to decreased time in the infusion room and it would decrease overall cost of care.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Female subjects must be either postmenopausal for at least 1 year before the screening visit, is surgically sterilized or if they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of SQ VELCADE, or agree to completely abstain from heterosexual intercourse.
* Male subjects, even if surgically sterilized must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse.
* Adults (age 18 to 80) with AML, excluding the M3 subtype, that are not likely to respond to conventional therapy
* Bone marrow and peripheral blood studies must be available for confirmation of diagnosis.
* Performance status of 60% or greater by the Karnofsky scale
* A minimum of 4 weeks must have elapsed since the completion of prior chemotherapy.
* Patients may have had autologous transplant.
* There are no minimum hematological parameter requirements prior to the first two cycles, as patients with AML and myelodysplastic syndrome (MDS) are understood to have low absolute neutrophil count (ANC) and platelet counts when the disease is active. However, patients with white blood cell count (WBC) greater than 30,000 will receive hydroxyurea to reduce the WBC count to below 30,000 at which point they may begin treatment.
* A pretreatment calculated creatinine clearance (absolute value) of ≥ 40 ml/minute or serum creatinine of < 1.5 x upper limit of normal is required.
* Patients must have a serum bilirubin ≤1.5 mg/dl, serum glutamic-oxaloacetic transaminase (SGOT) and serum glutamic-pyruvic transaminase (SGPT) ≤2.5 times the institutional upper limits of normal.

Exclusion Criteria:

* There is no specific platelet and absolute neutrophil count that will exclude patients from this study given the natural history of AML.
* Patient has greater than or equal to Grade 2 peripheral neuropathy
* Patient had myocardial infarction within 6 months prior to enrollment or has New York Heart Association Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant. An left ventricular ejection fraction (LVEF) must be > 50
* Patient has hypersensitivity to VELCADE, boron, or mannitol.
* Female subject is pregnant or lactating.
* Female patients who are lactating or have a positive serum pregnancy test during the screening period, or a positive urine pregnancy test on Day 1 before first dose of study drug, if applicable.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
* Radiation therapy within 3 weeks before randomization. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.
* Patients with active/uncontrolled central nervous system (CNS) leukemia
* Patients eligible, at the time of starting treatment, for curative therapeutic approaches (such as allogeneic transplant) are not eligible for the trial.
* Patients may not receive any other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) while on this study other than hydroxyurea for control of counts.
* Human Immunodeficiency Virus (HIV)-positive.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-12-19 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tuscano, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Comprehensive Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bortezomib + Doxil
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib + Doxil
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: The time from first day of treatment to the first observation of disease progression or death due to any cause. If a patient has not progressed or died, progression-free survival is censored at the time of last follow-up.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bortezomib + Doxil
Number analyzed (Participants) | 10
days | 21 [17 to NA] — Upper value of the confidence interval was not reached.

2. Secondary Outcome: Overall Survival
Description: Overall survival wil be measured as the time from start of treatment to the Date of death or the last date the patient was known to be alive
Time Frame: Up to two years
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Bortezomib + Doxil
Number analyzed (Participants) | 10
Days | 50 [41 to NA] — Upper value of the confidence interval was not reached.

3. Secondary Outcome: Toxicity Information Recorded Will Include the Type, Severity, Time of Onset, Time of Resolution, and the Probable Association With the Study Regimen.
Description: Toxicity will be evaluated based on the standard NCI Common Toxicity Criteria for Adverse Effects CTCAE) V.4.0 grading criteria.
Time Frame: Up to two years
Measure: Number; unit: participants
Arm/Group | Bortezomib + Doxil
Number analyzed (Participants) | 25
participants
  Abdominal pain | 4
  Alanine aminotransferase increased | 3
  Anemia | 17
  Anorexia | 7
  Aspartate aminotransferase increased | 4
  Chills | 4
  Constipation | 4
  Cough | 4
  Diarrhea | 9
  Dizziness | 8
  Dyspnea | 10
  Edema limbs | 3
  Epitaxis | 4
  Fatigue | 15
  Febrile neutopenia | 12
  Gastrointestinal disorders - Other, gum tenderness | 3
  Generalized muscle weakness | 4
  Headache | 5
  Hypoalbuminemia | 6
  Hypocalcemia | 4
  Hypokalemia | 3
  Hyponatremia | 7
  Hypotension | 4
  Infections and infestations - Other, bacteremia | 3
  Insomnia | 4
  Lymphocyte count decreased | 12
  Malaise | 4
  Mucositis oral | 4
  Nausea | 15
  Neutrophil count decreased | 10
  Peripheral sensory neuropathy | 4
  Platelet count decreased | 18
  Respiratory, thoracic and mediastinal disorders - Other, tachypnea | 3
  Skin and subcutaneous tissue disorders - Other, Ecchymoses | 4
  Vomiting | 8
  White blood cell decreased | 14

ADVERSE EVENTS:
Time Frame: Up to 30 days after discontinuation of study drugs.
Description: Incidence of adverse events.
Arm/Group | Bortezomib + Doxil
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 10/25
Other Adverse Events (participants affected / at risk) | 18/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib + Doxil (N=25)
Atrial fibrillation (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bronchial infection (Infections and infestations) | 1
bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Catheter related infection (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Heart failure (Cardiac disorders) | 1
Infections and infestations - Other, Bacteremia (Infections and infestations) | 1
neoplasms benign, malignant and unspecified (incl cysts and polyps) - other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Vasovagal reaction (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib + Doxil (N=25)
Abdominal pain (Gastrointestinal disorders) | 4
Alanine aminotransferase increased (Investigations) | 3
Anemia (Blood and lymphatic system disorders) | 17
Anorexia (Metabolism and nutrition disorders) | 7
Aspartate aminotransferase increased (Investigations) | 4
Bloating (Gastrointestinal disorders) | 2
Blood bilirubin increased (Investigations) | 2
Bruising (Injury, poisoning and procedural complications) | 2
Catheter related infection (Infections and infestations) | 2
Chills (General disorders) | 4
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Creatinine increased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 9
Dizziness (Nervous system disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
Edema limbs (General disorders) | 3
Epitaxis (Respiratory, thoracic and mediastinal disorders) | 4
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 15
Febrile neutropenia (Blood and lymphatic system disorders) | 12
Fever (General disorders) | 2
Gastrointestinal disorders - Other, Gum tenderness (Gastrointestinal disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 5
Heart failure (Cardiac disorders) | 2
Hematoma (Vascular disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 4
hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Insomnia (Psychiatric disorders) | 4
Lethargy (Nervous system disorders) | 2
Lymphocyte count decreased (Investigations) | 12
Malaise (General disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other: body/pain sore (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 15
neutrophil count decreased (Investigations) | 10
Pain (General disorders) | 2
Pain extremity (Musculoskeletal and connective tissue disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 4
Platelet count decreased (Investigations) | 18
presyncope (Nervous system disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory, thoracic and mediastinal disorders - Other, specify: Tachypnea (Respiratory, thoracic and mediastinal disorders) | 3
Sinus tachycardia (Cardiac disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify: Ecchymoses (Skin and subcutaneous tissue disorders) | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 8
Weight gain (Investigations) | 2
Weight loss (Investigations) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
White blood cell decreased (Investigations) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT01736943/Prot_SAP_000.pdf